CLINICAL TRIAL: NCT05588674
Title: Investigating a Novel Multi-strain Probiotic Supplement on Indices of Exercise Performance and Recovery
Brief Title: The Effect of Probiotics on Exercise Performance and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Biopolis S.L. (Industry)
Responsible Party: Principal Investigator, Liam Heaney, Senior Lecturer/Principal Investigator, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LEON7551
Record Dates: First submitted 2022-10-01; First posted 2022-10-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-02

CONDITIONS: Probiotics; Acute Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic Supplement (Experimental): 1 billion CFU per capsule of a multistrain probiotic formulation including one Bifidobacterium and two Lactobacilli strains with maltodextrin as a carrier
  Interventions: Dietary Supplement: Probiotic Supplement
- Placebo capsule (Placebo Comparator): 418mg maltodextrin
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Probiotic Supplement — 8.5 week supplementation period. One capsule daily.
  Arms: Probiotic Supplement
Other: Placebo Capsule — 8.5 week supplementation period. One capsule daily.
  Arms: Placebo capsule

SUMMARY:
This project will involve administering a multi-strain probiotic supplement to investigate the capacity to improve exercise performance and/or recovery. This will be done by assessing physiological measures (e.g. performance and muscle soreness), biochemical measures (e.g. oxidative stress and inflammation), and microbial diversity (i.e. associations with bacteria present in the gut). Participants will be well-trained, recreational exercisers and will visit the laboratory a total of eight times, including an 8-week probiotic vs placebo supplementation period.

DETAILED DESCRIPTION:
A total of 36 healthy, and active men and women aged 18-40 years of age will be recruited and allocated randomly into either a probiotic or placebo group, where both the investigator and participants will be blinded to the supplements (double-blind randomised control trial format).

Each participant will be asked to attend the research laboratory on eight separate occasions and to refrain from high-intensity exercise (e.g. long-distance running, competitive sport, weightlifting) in the 48 hours prior to each visit and light exercise (e.g. mild jogging or long walk) the day before each visit. They will also be asked to refrain from alcohol intake for 24 hours before each visit and caffeine intake on the morning of the visit.

Visit 1

Following consent, the participants will complete a ramp incremental exercise test for determination of volume of peak oxygen uptake (VO2peak) and the first abrupt change in the oxygen (VO2) and carbon dioxide (VCO2) concentrations of the expired air known as Gas Exchange Threshold (GET). The data collected during the incremental test will be used to calculate the work rates which will be employed during the subsequent exercise tests. The participant will also be asked to complete a food frequency and exercise questionnaire to understand general dietary and training practices.

Visit2

At least 48 hours following visit 1, the participant will return to the exercise laboratory in the morning after a 10-hour overnight fast, where they will complete a familiarisation to the cycling time trial performance test. The time trial will consist of a short 10 min warm-up cycle at the power output equivalent to 95% GET followed by a partial time trial of fixed work at self-selected cycling speed and a full time trial of fixed work at self-selected cycling speed. The participant will also be shown a demonstration for the use of a faecal collection sampling device that will be used prior to the following visit, the device will be given to them to take away from the laboratory at used at home.

Visit 3

At least 72 hours hours following visit 2, the participant will be asked to attend the laboratory during the morning of the trial after after a 10-hour overnight fast. Participants will then complete visual analogue scales (VAS) to assess their appetite ratings. Appetite ratings will be assessed using 100 m VAS. They will then be provided with a standardised breakfast. The participant will also be asked to collect faecal samples at any convenient point in the 48 hours prior to the visit. The participant will then complete a questionnaire to assess their mood and anxiety profile as well as a food frequency questionnaire (FFQ). Other routine anthropometric information will be collected including height, body mass, blood pressure/pulse wave analysis, resting heart rate, body fat % and lean body mass, following a resting period. The participant will complete an exercise protocol that consists of a 45 min steady-state exercise at 95% GET intensity calculated from familiarisation trial. Following completion of the steady-state exercise, the participant will be asked to complete a cycling performance time trial in which they will be asked to complete a set amount of work as quickly as they are able. The work target is estimated using data obtained during familiarisation time trial. The set workload will be adjusted for female participants. Blood sampling will be collected prior to and following the steady-state exercise, and following completion of the time trial. Participants will then be randomised into a study group (probiotic or placebo). The participant will be asked to take the first dose prior to leaving the laboratory, with further doses of one capsule per day with breakfast.

Visit 4

During week 7 of supplementation, the participant will return to the laboratory to repeat the time trial completed as part of experimental trial 1 as a re-familiarisation exercise. Participants will then be familiarised with performing a counter movement jumps (CMJ). Thereafter, they will be familiarised with a hand-held pressure pain threshold (PPT) algometer.

Visit 5

Following 8 weeks from visit 3, the participants will return to the laboratory at after a 10-hour overnight fast. They will provide faecal samples (collected within 48 hours prior to the visit) and complete appetite, mood and anxiety questionnaires alongside a repeat FFQ. They will then repeat the same exercise performance testing protocol as done in Visit 3. Following the cessation of the performance trial 2, the participant will rest for at least 15 minutes or until their heart rate has returned to within 30 bpm of their pre-exercise level. They will then complete 100 drop jumps. Blood sampling will be collected prior to and following the steady-state exercise, following completion of the time trial, and at 1-hour after the completion of the drop jumps.

Visits 6, 7 and 8

The participant will be asked to return to the laboratory at 24, 48 and 72 hours post-Visit 5 after a 10-hour overnight fast and a resting blood sample will be collected. Subsequently, participants will perform 3 CMJs, 30 s apart with passive recovery. Then they will be asked to perform a squat and then rate their current delayed onset muscle soreness (DOMS) using a 200 mm (VAS) for generalised muscle pain. A hand-held PPT algometer will be used for the assessment of muscle-specific soreness at specific sites across the major muscles groups of the lower limbs. All sites will be marked to ensure that pressure is applied at the same spot for each repetition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Involved in regular or structured exercise/sport programmes

Exclusion Criteria:

* Current use or previous use within 3 months of probiotic supplements
* Current use or previous use within 3 months of antibiotics
* A recent history of surgery/injury associated with impairment of cycling performance
* History of chronic disease (excluding mild asthma)
* Poor tolerance to any component of the supplement
* Any blood-borne disorder/disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Exercise Performance | 8 weeks
  Pre- and post-supplementation levels of exercise performance tested via a cycle ergometer time trial
Functional Exercise Recovery | 4 days
  Assessment of recovery from muscle damaging exercise through the measurement of pre- and post-damaging exercise testing of counter movement jump height
Recovery from Muscle Soreness | 4 days
  Assessment of recovery from muscle damaging exercise through the measurement of pre- and post-damaging exercise testing of muscle soreness using VAS scales and handheld pain threshold algometer
Biochemical Recovery from Exercise (Inflammation) | 4 days
  Assessment of recovery from muscle damaging exercise through the measurement of pre- and post-damaging exercise testing of inflammatory markers (IL-6, CRP) by immunoassay
Biochemical Recovery from Exercise (Tissue Damage) | 4 days
  Assessment of recovery from muscle damaging exercise through the measurement of pre- and post-damaging exercise testing of markers of muscle damage (CK, LDH) by immunoassay
Biochemical Recovery from Exercise (Oxidative Stress) | 4 days
  Assessment of recovery from muscle damaging exercise through the measurement of pre- and post-damaging exercise testing of markers of oxidative stress (8-OHDG, MDA) by immunoassay

SECONDARY OUTCOMES:
Gut Microbial Diversity Testing by 16S Sequencing | 8 weeks
  Assessment of gut microbial diversity pre- and post-supplementation via faecal sampling

CONTACTS AND LOCATIONS:
Overall Officials: Liam M Heaney, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No